CLINICAL TRIAL: NCT06698887
Title: Long-Term Safety Follow-Up Surveillance for Phase 3 Trial (KarMMA-9/CA089-1043) to Compare the Efficacy and Safety of Idecabtagene Vicleucel With Lenalidomide Maintenance Therapy Versus Lenalidomide Maintenance Therapy Alone in Adult Participants With Newly Diagnosed Multiple Myeloma Who Have Suboptimal Response After Autologous Stem Cell Transplantation
Brief Title: A Study to Evaluate the Long-Term Safety of Idecabtagene Vicleucel Treatment in Adults With Newly Diagnosed Multiple Myeloma in Korea
Status: Recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA089-1081
Record Dates: First submitted 2024-11-19; First posted 2024-11-21 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — idecabtagene vicleucel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants receiving idecabtagene vicleucel
  Interventions: Drug: Idecabtagene vicleucel

INTERVENTIONS:
Drug: Idecabtagene vicleucel — As per CA089-1043 study protocol

SUMMARY:
The purpose of this study is to monitor the long-term safety of participants who received idecabtagene vicleucel treatment as part of the KarMMa-9 (CA089-1043) Phase 3 clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants ≥19 years of age
* Korean participants with newly diagnosed multiple myeloma who had a suboptimal response after autologous stem cell transplantation (ASCT) and who were treated with idecabtagene vicleucel (assigned to Arm A) in the KarMMa-9 trial (CA089-1043)
* Participants must understand and voluntarily sign and informed consent form (ICF) for the Korea long-term follow-up surveillance study prior to any surveillance-related procedures being conducted

Exclusion Criteria:

* Participants who participate in KarMMa-9 trial (CA089-1043) but disagree with long-term follow-up surveillance in Korea
* Participants who are not possible to treat with Ide-cel within 9 days post-completion of lymphodepleting chemotherapy (LDC), if delays occur. However, depending on the participants recovery status, whether idecabtagene vicleucel is administered or not, should be discussed with a medical monitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with newly diagnosed multiple myeloma (NDMM) who had a suboptimal response after autologous stem cell transplantation (ASCT) and who were treated with idecabtagene vicleucel in the KarMMa-9 (CA089-1043) Phase 3 clinical trial.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2031-03-27 (Estimated); Study Completion 2031-03-27 (Estimated)

PRIMARY OUTCOMES:
Participant adverse events | Monthly from months 4-18, every 2 months from months 19-59, and annually from month year 5 to 15
Number of participants with positive replication-competent lentivirus test results | At 4, 7, 13, and 25 months, and annually up to 15 years
Persistent vector sequence monitoring | Months 7-18 and annually from years 5-15

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Monthly up to 18 months and every two months after month 19 up to 15 years
Overall survival (OS) | Every 3 months up to month 60, annually thereafter up to 15 years
Number of participants that achieve complete response or stringent complete response | At months 4-18, every 2 months from months 19-59, and annually from years 5-15
Health-related quality of life (HRQoL) measured by the European Organization for Research and Treatment of Cancer core quality of life (EORTC QLQ-C30) questionnaire | At months 4-18, every 2 months from months 19-59, and annually from years 5-15
Health-related quality of life (HRQoL) measured by the European Organization for Research and Treatment of Cancer assessment of quality of life of myeloma patients (EORTC QLQ-MY20) questionnaire | At months 4-18, every 2 months from months 19-59, and annually from years 5-15
Health-related quality of life (HRQoL) measured by the EuroQol-5 Dimensions-5 Levels (EQ-5D-5L) questionnaire | At months 4-18, every 2 months from months 19-59, and annually from years 5-15

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (5):
- South Korea (5):
  - Chonnam National University Hwasun Hospital, Hwasun, Jeonranamdo
  - Seoul National University Hospital, Seoul, Seoul-teukbyeolsi [Seoul]
  - Asan Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
  - Samsung Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
  - The Catholic Univ. of Korea Seoul St. Mary's Hospital, Seoul, Seoul-teukbyeolsi [Seoul]

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts